CLINICAL TRIAL: NCT04487327
Title: The Effect of Needle Placement on Muscle Stiffness, Gait, Balance, Pain and Functional
Brief Title: The Effect of Needle Placement on Muscle Stiffness, Gait, Balance, Pain and Functional Outcomes in Individuals With Injury to the Ankle and/or Hindfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Principal Investigator, Stephanie Albin, Principal Investigator, Regis University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: albin2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-27 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Ankle and or Hindfoot Injury
Keywords: dry needling; muscle stiffness; ankle injury; hindfoot injury; plantar pressure
MeSH Terms: conditions — Ankle Injuries | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Specific Aim 1: To evaluate if DN has an effect on muscle stiffness, gait, pain pressure threshold, and balance in individuals with injuries to the ankle and/or hindfoot.
  The dependent variables for Aim1 are: muscle stiffness, plantar pressure, PPT, and balance. The independent variables for Aim1 are Group (MTrP needling versus away from the MTrP site) and Time. The primary aim will be examined using linear mixed modeling with any baseline differences between groups used as a co-variate. A separate model will be created for each dependent variable.
  Specific Aim 2: To determine the validity of dry needling specific muscles of the lower extremity based upon needle placement, location relative to anatomical structures and accuracy of needle placement in muscle with in vivo ultrasound imaging.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study investigators collecting outcome assessments will be blinded to group allocation. Participants will be asked not to reveal what group they believe they were randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling within the Myofascial Trigger Point (Experimental): Randomized to receive DN at the site of the MTrP
  Interventions: Other: Dry Needling
- Dry Needling away from Myofascial Trigger Point Site (Active Comparator): Randomized to receive DN 2 cm away from the site of the MTrP but within the same muscle
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — The dry-needling treatment will consist of inserting a sterile needle into 2-4 muscles of the participant either at the MTrP or 2 cm away from the MTrP, but within the same muscle. To assist in the reduction of infection risk and protection of the participants, the site will be cleaned with alcohol prior to treatment and investigators performing the needling treatment will wear gloves and handle needles using aseptic technique throughout the procedure. Each needle insertion will last approximately 5 seconds using a "pistoning" (in and out) technique.

SUMMARY:
The purpose of this randomized controlled trial is to assess the effect of DN at either the site of the identified myofascial trigger point/s (MTrP) of in the same muscle, but away from the MTrP site/s in individuals with ankle and/or hindfoot injury. Assessments will be of self-reported outcomes, self-reported pain, gait, balance, muscle stiffness, and pain pressure threshold. The secondary purpose of this study is to determine the validity of dry needling specific muscles of the lower extremity based upon needle placement, location relative to anatomical structures and accuracy of needle placement in muscle using ultrasound imaging.

DETAILED DESCRIPTION:
Few studies have assessed the validity of needling muscles of the lower extremity. For muscles such as the tibialis posterior that are not easily accessible or directly palpable secondary to the deep anatomical position and due to the proximity of the tibial nerve and the posterior tibial artery within the deep compartment, examining accurate needle placement is clinically relevant. In addition, DN has been shown to be a beneficial management strategy for individuals with lower extremity condition; however, the investigators may be able to optimize these beneficial effects by performing DN on the MTrP versus other sites within the same muscle.

If needling directly into the MTrP is more effective than needling away from the MTrP but into the same muscle, it is possible that the improved efficiency could help to optimize management of patients with injury to the ankle/hindfoot with less visits and potentially decreasing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a previous lower extremity injury occurring to the ankle and/or hindfoot within the previous 12 months AND
* pain greater than 3 out of 10 on the numeric pain rating scale (NPRS) OR
* limited weightbearing dorsiflexion range of motion of greater than 2.0 cm side-to-side difference as measured by the ankle lunge test (ALT) OR
* greater than 3.5% side-to-side difference as assessed by the Y-balance test.

Exclusion Criteria:

* Operative fixation within the past 3 months to the lower extremity
* Have received DN of the lower extremity within the past 30 days
* Current pregnancy
* Have a history of systemic disorders in which DN would be contraindicated (bleeding disorders or current anticoagulant medication use)
* Immunocompromised
* Decline participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
DN location effect on self-reported and clinical outcomes | 2 year
  Foot and Ankle Ability Measure (FAAM)
DN location effect on clinical outcomes - Muscle Stiffness | 2 year
  Muscle Stiffness Measured with the MyotonPro
DN location effect on clinical outcomes - Gait | 2 year
  Plantar pressure during gait measured by the EMED system and GAITRite
DN location effect on clinical outcomes - Dynamic Balance | 2 year
  Balance measured by the Y-balance test
DN location effect on clinical outcomes - PPT | 2 year
  Pain pressure threshold measured by an algometer

SECONDARY OUTCOMES:
Validation of needle placement in lower extremity muscles | 6 month
  Individuals will receive dry needling with the aseptic technique previously described. With the needle in place, diagnostic ultrasound will be performed. The accuracy of the needle placement will be assessed and the distance from the needle to major arteries, nerve, and veins will be measured in millimeters and documented. Only one visit lasting approximately 30 minutes will be required for this portion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Albin, Principal Investigator — Regis University
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pecos-Martin D, Montanez-Aguilera FJ, Gallego-Izquierdo T, Urraca-Gesto A, Gomez-Conesa A, Romero-Franco N, Plaza-Manzano G. Effectiveness of dry needling on the lower trapezius in patients with mechanical neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2015 May;96(5):775-81. doi: 10.1016/j.apmr.2014.12.016. Epub 2015 Jan 9. PMID 25582412
- [Background] Fernandez-de-Las-Penas C, Mesa-Jimenez JA, Paredes-Mancilla JA, Koppenhaver SL, Fernandez-Carnero S. Cadaveric and Ultrasonographic Validation of Needling Placement in the Cervical Multifidus Muscle. J Manipulative Physiol Ther. 2017 Jun;40(5):365-370. doi: 10.1016/j.jmpt.2017.03.002. Epub 2017 Apr 13. PMID 28413118